CLINICAL TRIAL: NCT02800187
Title: The Effect of Extracorporeal Shock Wave Therapy in Patients With Mild to Moderate Carpal Tunnel Syndrome
Brief Title: The Dose Effect of Extracorporeal Shock Wave Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Physical medicine and rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 2-105-05-031
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- three-sessions of ESWT (Experimental): Active three-sessions of ESWT ( once a week for 3 weeks) was given.
  Interventions: Device: ESWT
- one-session of ESWT (Active Comparator): One-session of ESWTactive ESWT was given.
  Interventions: Device: ESWT
- Night splint (Active Comparator): The night splint was firmly fixed in a neutral position to immobilize the affected wrist. Patients were ordered to wear the splint while resting at night and at least 8 hours per day during the period of study. Another 3 sessions of sham ESWT was given.
  Interventions: Device: ESWT

INTERVENTIONS:
Device: ESWT — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs).

SUMMARY:
The shock wave is a new and potential intervention for the reinnervation of peripheral nerve. The purpose of this study was to assess the dose effect of extracorporeal shock wave therapy on carpal tunnel syndrome.

DETAILED DESCRIPTION:
The investigator perform a prospective randomized, single-blinded study to investigate the dose effect of ESWT in patients with carpal tunnel syndrome.

The evaluation was performed pretreatment as well as on the 4th, 8th, 12th, 16th and 24 week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 year-old.
2. Typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test, numbness/tingling in at least two of the first, second, or third digits, and in whom the diagnosis was confirmed using an electrophysiological study.

Exclusion Criteria:

1. Cancer
2. Coagulopathy
3. Pregnancy
4. Inflammation status
5. Patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previously undergone wrist surgery or steroid injection for CTS.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline of cross-sectional area in median nerve on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline of electrophysiological study on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  electrophysiological study according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wu YT, Ke MJ, Chou YC, Chang CY, Lin CY, Li TY, Shih FM, Chen LC. Effect of radial shock wave therapy for carpal tunnel syndrome: A prospective randomized, double-blind, placebo-controlled trial. J Orthop Res. 2016 Jun;34(6):977-84. doi: 10.1002/jor.23113. Epub 2015 Dec 10. PMID 26610183
- [Result] Seok H, Kim SH. The effectiveness of extracorporeal shock wave therapy vs. local steroid injection for management of carpal tunnel syndrome: a randomized controlled trial. Am J Phys Med Rehabil. 2013 Apr;92(4):327-34. doi: 10.1097/PHM.0b013e31826edc7b. PMID 23044704